CLINICAL TRIAL: NCT06289985
Title: STEP: StrokeNet Thrombectomy Endovascular Platform
Brief Title: StrokeNet Thrombectomy Endovascular Platform
Acronym: STEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Cincinnati (Other); University of Virginia (Other); Berry Consultants (Other); University of California, Los Angeles (Other); MOUNT SINAI HOSPITAL (Other); The Cooper Health System (Other); University of Pittsburgh Medical Center (Other); Stony Brook University (Other); University at Buffalo (Other)
Responsible Party: Principal Investigator, Jordan Elm, Research Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: STEP; 1OT2NS129366-01 (NIH)
Record Dates: First submitted 2024-02-13; First posted 2024-03-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Practice Management, Medical

STUDY DESIGN:
Intervention Model Description: Adaptive Bayesian Platform Trial evaluating multiple interventions in multiple domains.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Endovascular Therapy (EVT) Indication Expansion Domain: Low NIHSS Strata (Other): Adult patients with acute cerebral ischemia within 24 hours of last known well who have large vessel occlusion (LVO) and mild deficits/low NIHSS (NIHSS 0-5) will be randomized to receive one of two strategies:
  * Endovascular Therapy (EVT)
  * Medical Management (MM)
  Interventions: Device: Endovascular thrombectomy with any FDA-approved category POL or NRY device; Other: Medical Management
- Endovascular Therapy (EVT) Indication Expansion Domain: Medium/Distal Occlusions Strata (Other): Adult patients with acute cerebral ischemia within 24 hours of last known who have Medium Vessel Occlusion (MVO) with Non-dominant/Co-dominant M2 occlusion or Distal Medium Vessel Occlusion (DMVO) patients with M3 occlusion will be randomized to receive one of two strategies:
  * Endovascular Therapy (EVT)
  * Medical Management (MM)
  Interventions: Device: Endovascular thrombectomy with any FDA-approved category POL or NRY device; Other: Medical Management

INTERVENTIONS:
Device: Endovascular thrombectomy with any FDA-approved category POL or NRY device — Endovascular thrombectomy with any FDA-approved category POL or NRY device - Neurovascular Mechanical Thrombectomy Device For Acute Ischemic Stroke Treatment (POL), and/or Catheter, Thrombus Retriever (NRY)
  Other Names: EVT; Endovascular Recanalization Therapy; Endovascular Therapy
Other: Medical Management — Medical Management (MM) may involve any combination of the following: intravenous thrombolysis, antiplatelets, anti-hypertensives, cholesterol-lowering medications, and rehabilitative care.

SUMMARY:
STEP is a Randomized, Multifactorial, Adaptive Platform trial that seeks to optimize the care of patients with acute ischemic stroke (AIS) due to large (LVO) or medium vessel occlusions (MVO).

DETAILED DESCRIPTION:
The StrokeNet Thrombectomy Endovascular Platform (STEP) is conducted within NIH StrokeNet at 38 comprehensive stroke centers across the US. The primary goal is to optimize all aspects of care of acute ischemic stroke patients with a large or a medium vessel occlusion. The platform trial operates under an overarching Master Protocol in an inferentially integrated framework. The platform trial is designed to support the studies of three broad categories of therapeutics: expansion of endovascular treatment (EVT) indications, innovative EVT devices and concomitant medical therapies, and novel pre- and early-hospital technologies and systems of care. As new interventions are put forth, they will be added to the Master Protocol as a new Domain or part of an existing Domain. STEP utilizes a flexible Bayesian design with frequent adaptive analyses to assess whether a given intervention is superior, inferior, or equivalent either within a Domain or for specific populations within the Domain.

ELIGIBILITY:
STEP PLATFORM INCLUSION CRITERIA:

1. Suspected diagnosis acute ischemic stroke
2. Likely causative intracranial large or medium vessel occlusion

STEP PLATFORM EXCLUSION CRITERIA:

1. Proven contraindication to endovascular thrombectomy
2. Prisoners/incarcerated

DOMAIN-SPECIFIC ELIGIBILITY CRITERIA:

Each domain may have additional eligibility criteria.

STEP EVT INDICATION EXPANSION DOMAIN INCLUSION CRITERIA:

1. Age 18 years or older 2. Pre-stroke modified Rankin Scale score 0-2 3. Presentation to enrolling hospital within 24 hours of last known well/stroke onset 4. Able to initiate arterial puncture within 2 hours from qualifying CTA/MRA or CTP/MRP imaging

*CT/MR and qualifying CTA/MRA or CTP/MRP should be repeated if more than 120 minutes have elapsed since the imaging and randomization has not been performed. The exception is for LVO Mild deficit/Low NIHSS 0-5 for which imaging would only need to be repeated if there has been significant improvement in the NIHSS prior to randomization.

5. Has one of the following presentations:

1. LVO patients with mild deficits/low NIHSS (must have both):

   1. Mild presenting neurologic deficits - NIHSS 0-5 (Must have some focal neurological deficit attributable to the target occlusion if NIHSS 0)
   2. Complete occlusion of the intracranial Internal Carotid Artery (ICA) or M1 Middle Cerebral Artery (MCA)
2. Medium/Distal Vessel Occlusion:

   1. Visualized complete occlusion or perfusion deficit (Tmax > 4s) supportive of a cortical branch occlusion in one of the following vessels:

      i) Non-dominant/Co-dominant M2 (defined as serving < 50% of entire overall MCA territory) ii) M3
   2. If symptom onset is > 6h, the core must be less than 50% of the territory supplied by the occluded vessel as evident by either:

      i) Hypodensity and loss of grey-white border on NCCT or ii)ADC <620 mm2/s on diffusion MRI or rCBF<30% on CTP
   3. NIHSS > =8

STEP EVT INDICATION EXPANSION DOMAIN EXCLUSION CRITERIA:

1. Clinical

   1. Presumed septic embolus; suspicion of bacterial endocarditis
   2. Seizure at stroke onset or between onset and enrollment
   3. Known anaphylactic reaction to contrast material that precludes endovascular reperfusion therapy
   4. Intracranial occlusion suspected to be chronic, based on history and/or imaging
   5. Intracranial dissection, based on history and/or imaging
   6. Cerebral vasculitis, based on history and/or imaging
   7. Known pregnancy
   8. Known pre-existing medical, neurological or psychiatric disease that would confound the neurological or functional evaluations
   9. Known serious, advanced, or terminal illness or life expectancy less than 6 months in the investigator judgment
   10. Known or high suspicion for underlying intracranial atherosclerotic disease (ICAD)
2. Laboratory

   a. Known platelet count <100,000/uL
3. Imaging

   1. CT ASPECT score <6 (MRI ASPECT score <7)
   2. Unfavorable vascular anatomy that limits access to the occluded artery precluding endovascular reperfusion therapy.
   3. Acute occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation)
   4. Tandem occlusions
   5. Significant mass effect with midline shift (>5mm)
   6. Evidence of intra-cranial tumor (except small meningioma defined as (1) <=3 cm, (2) asymptomatic) as confirmed on CT/MRI)
   7. Evidence of acute intracranial hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Global disability measured by Modified Rankin Score | 90-day
  The modified Rankin Score is a 7-outcome ordinal scale where 0 = No symptoms and 6= Dead.
  The analysis of the primary endpoint will be based on a utility weighting of the 7 outcomes, where 0 represents the worst possible health state and 1 represents the best possible state.

OTHER OUTCOMES:
Global disability measured by Modified Rankin Score | 1 day of hospital discharge
  The modified Rankin Score is a 7-outcome ordinal scale where 0 = No symptoms and 6= Dead.
Neurological deficit as measured by the National Institutes of Health Stroke Scale (NIHSS) | 24 (+/-12) hours after the time of randomization
  NIHSS is a stroke severity score that ranges from 0 to 42, with higher numbers indicating a more severe stroke.
Symptomatic intracranial hemorrhage | 36 hours after randomization
  modified Heidelberg definition
Any radiologic intracranial hemorrhage | 36 hours after randomization
  any acute intracranial blood, symptomatic or asymptomatic
Mortality | 90 days
  all cause deaths

CONTACTS AND LOCATIONS:
Overall Officials: Jordan J Elm, PhD, Principal Investigator — Medical University of South Carolina; Eva A Mistry, MBBS, MSCI, Principal Investigator — University of Cincinnati; Pooja Khatri, MD, Principal Investigator — University of Cincinnati; Colin P Derdeyn, MD, Principal Investigator — University of Virginia; Jeffery L Saver, MD, Principal Investigator — University of California, Los Angeles; Tudor G Jovin, MD, Principal Investigator — The Cooper Health System; Raul G Nogueira, MD, FAHA, Principal Investigator — University of Pittsburgh; David Fiorella, MD, PhD, Principal Investigator — Stony Brook University; Adnan Siddiqui, MD, PhD, Principal Investigator — University at Buffalo; J Mocco, MD, MS, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (41):
- United States (41):
  - University of Alabama Hospital, Birmingham, Alabama
  - UCSD Health La Jolla, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCSD Medical Center - Hillcrest Hospital, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Jackson Memorial Hospital, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - M Health Fairview Southdale Hospital, Edina, Minnesota
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - Barnes Jewish Hospital, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - NYU Langone Hospital, Brooklyn, New York
  - Buffalo General Medical Center, Buffalo, New York
  - The Mount Sinai Hospital, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - UH Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC Mercy Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina University Hospital, Charleston, South Carolina
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Medical City Plano, Plano, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Utah Healthcare, Salt Lake City, Utah
  - UVA Medical Center, Charlottesville, Virginia
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level case report form data will be made available for research purposes upon completion of the trial. Low incidence values and free text fields will be collapsed or removed to ensure participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after study is completed.
Access Criteria: NIH/NINDS website